CLINICAL TRIAL: NCT01121250
Title: Spouse READI (Resilience Education And Deployment Information) Post Deployment Telephone Support Groups
Acronym: Spouse READI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memphis VA Medical Center (U.S. Federal Agency)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Linda O. Nichols, Ph.D., Healthcare education specialist/Health Services Researcher, Memphis VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: W81XWH-09-1-0242
Record Dates: First submitted 2010-05-07; First posted 2010-05-12 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-10

CONDITIONS: Spouses; Military Personnel; Coping Skills
Keywords: Combat disorders; Spouses; Support; Military personnel
MeSH Terms: conditions — Combat Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telephone Discussion Groups (Experimental): Each telephone discussion group will meet 12 times during six months. The one-hour calls will be semi-structured conference calls with education, training in coping skills and cognitive restructuring, and support. A Participant Workbook will include comprehensive materials for all sessions and topics, other resources, and red flag resources - areas that may exacerbate problems, add a level of difficulty or distress, and/or indicate a need for referrals (e.g., unsafe behaviors, substance abuse, spouse abuse, PTSD, depression, traumatic brain injury).
  Interventions: Behavioral: Telephone Discussion Groups
- Education sessions (Active Comparator): Participants will have 12 sessions (delivered using slides and telephone) that cover the same education content, without skills building or support, over six months. They will also receive the Participant Workbook.
  Interventions: Behavioral: Education sessions
- Usual Care (No Intervention): Participants do not receive any services.

INTERVENTIONS:
Behavioral: Telephone Discussion Groups — Each telephone discussion group will meet 12 times during six months. The one-hour calls will be semi-structured conference calls with education, training in coping skills and cognitive restructuring, and support. A Participant Workbook will include comprehensive materials for all sessions and topics, other resources, and red flag resources - areas that may exacerbate problems, add a level of difficulty or distress, and/or indicate a need for referrals (e.g., unsafe behaviors, substance abuse, spouse abuse, PTSD, depression, traumatic brain injury).
  Arms: Telephone Discussion Groups
Behavioral: Education sessions — Participants will have 12 sessions (delivered using slides and telephone) that cover the same education content, without skills building or support, over six months. They will also receive the Participant Workbook.
  Arms: Education sessions

SUMMARY:
This 12-month study is for spouses or significant others of service members who have returned from Afghanistan or Iraq. This study will determine if participating in a telephone discussion group, offering education, skills building, and support, will help increase post-deployment adjustment. There will be 225 spouses recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

1. have a spouse who participated in a deployment to Iraq and Afghanistan and is at least 1 month post-deployment
2. if not married, must have lived as married for at least one year
3. must be committed to the relationship
4. have a telephone.

Exclusion Criteria:

1. known deployment of spouse in the next six months
2. auditory impairment that would make telephone use difficult.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2009-10; Primary Completion 2013-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda O Nichols, Ph.D., Principal Investigator — Memphis VA Medical Center and University of Tennessee Health Science Center; Jennifer L Martindale-Adams, Ed.D., Principal Investigator — University of Tennessee Health Science Center and VA Medical Center Memphis
Locations (1):
- Memphis VA Medical Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nichols, L.O., Martindale-Adams, J., Zuber, J., Graney, M., Burns, R., & Clark, C. Support for Spouses of Post Deployment Service Members. Military Behavioral Health, Published online: 30 Jan 2015. DOI:10.1080/21635781.2015.1009210
- [Result] Nichols L.O., Martindale-Adams, J., Zuber, J., & Graney, M. Service Member Need and Supportive Services Use of Military/Veteran Spouses. Military Behavioral Health, Published online: 09 Feb 2015, DOI:10.1080/21635781.2014.995251
- See also: Related Info — http://www.memphis.va.gov/spousesupport

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telephone Discussion Groups | Education Sessions | Usual Care
Started | 76 | 76 | 76
Completed | 76 | 76 | 75
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telephone Discussion Groups | Education Sessions | Usual Care | Total
Number analyzed (Participants) | 76 | 76 | 75 | 227
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (8.6) | 38.0 (8.3) | 35.1 (8.7) | 36.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 75 | 75 | 224
  Male | 2 | 1 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 10 | 27
  Not Hispanic or Latino | 66 | 69 | 65 | 200
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 3 | 4
  Asian | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 13 | 5 | 28
  White | 61 | 60 | 59 | 180
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 76 | 76 | 75 | 227

OUTCOME MEASURES:

1. Primary Outcome: Spouse Self-report of Anxiety
Description: Anxiety symptoms from the Generalized Anxiety Disorder-7 (GAD-7) scale, measured from 0-21, higher scores indicate greater anxiety
Time Frame: Baseline, 6 months, and 12 months
Population: All participants with anxiety data at baseline, six months, and twelve months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Discussion Groups | Education Sessions | Usual Care
Number analyzed (Participants) | 76 | 76 | 75
units on a scale
  Anxiety score at baseline | 7.9 (5.5) | 7.1 (5.1) | 7.9 (4.8)
  Anxiety score at 6 months | 5.5 (4.0) | 5.2 (4.4) | 6.2 (4.4)
  Anxiety score at 12 months | 6.0 (4.8) | 6.1 (4.9) | 5.5 (4.8)

2. Primary Outcome: Spouse Self-report of Depression
Description: Depression symptoms as measured on the Patient Health Questionnaire (PHQ-9), measured from 0-27, with higher numbers indicating more depression
Time Frame: Baseline, 6 months, and 12 months
Population: All participations with depression data at baseline, six and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Discussion Groups | Education Sessions | Usual Care
Number analyzed (Participants) | 76 | 76 | 75
units on a scale
  Depression symptoms at baseline | 6.6 (5.8) | 5.8 (5.2) | 6.4 (4.7)
  Depression symptoms at 6 months | 4.5 (4.6) | 4.4 (4.8) | 5.3 (4.1)
  Depression symptoms at 12 months | 4.8 (5.1) | 5.3 (4.8) | 5.0 (4.7)

3. Primary Outcome: Spouse Self-report of Resilience
Description: Resilience as measured on the Connor-Davidson Resilience Scale, measured from 0-100; higher scores show greater resilience
Time Frame: Baseline, 6 months, and 12 months
Population: All participants with resilience data at baseline, 6 and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Discussion Groups | Education Sessions | Usual Care
Number analyzed (Participants) | 76 | 76 | 75
units on a scale
  Resilience scores at baseline | 75.8 (10.0) | 78.8 (10.6) | 76.4 (9.5)
  Resilience scores at 6 months | 78.1 (12.4) | 77.9 (13.0) | 77.7 (10.7)
  Resilience scores at 12 months | 78.1 (11.0) | 76.3 (12.5) | 78.0 (10.2)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Telephone Discussion Groups | Education Sessions | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/76 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/76 | 0/75
Other Adverse Events (participants affected / at risk) | 0/76 | 0/76 | 0/75

LIMITATIONS AND CAVEATS:
Spouses were not screened for distress and did not exhibit high levels of anxiety or depression or low levels of resilience at baseline. Participants discontinued or were lost to follow up. Less than half of participants attended > six sessions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No